CLINICAL TRIAL: NCT05888805
Title: Myopia Control Efficacy of Second-generation DIMS Spectacle Lenses on Fast Progressing Myopes - Auxiliary Group
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: HOYA Lens Thailand LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0043588
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: Myopia; Defocus
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Participants will be prescribed with a pair of DIMS spectacle lenses for 24 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DIMS lens group (Other): Participants will be prescribed with a pair of DIMS spectacle lenses for 24 months.
  Interventions: Other: DIMS spectacle lens

INTERVENTIONS:
Other: DIMS spectacle lens — DIMS spectacle lens is a multifocal spectacle lens that corrects the distance refraction and provides myopic defocus simultaneously.
  Other Names: MiYOSMART

SUMMARY:
The purpose of this study is to examine the efficacy and performance of the Defocus Incorporated Multiple Segments (DIMS) Spectacle lenses on controlling myopia progression in fast progressing myopic children.

DETAILED DESCRIPTION:
DIMS spectacle lens is a multifocal spectacle lens that produces myopic defocus images and corrects distance refractive errors at the same time.

Participants will be prescribed a pair of DIMS spectacle lenses. Their cycloplegic refraction and axial length will be monitored every 6 months over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* SER: -1.00D or below
* Documented history of fast progressing myopia, either in SER or AL
* SER progression: 0.50D/year or more
* AL elongation: 0.27mm/year or more
* Best-corrected monocular visual acuity (VA) in both eyes: 0.00 logMAR (equivalent) or better
* Acceptance of random group allocation and the masked study design
* Anisometropia of 1.50 D or less
* Astigmatism of 2.00 D or less

Exclusion Criteria:

* Strabismus and binocular vision abnormalities
* Ocular and systemic abnormalities
* Prior experience of myopia control

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Estimated)
Dates: Start 2023-07-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refraction change in spherical equivalent refraction (SER) | Baseline, 1st year and 2nd year
  Cycloplegic SER (in diopter) will be measured using an open field autorefractor.
  Change in SER with cycloplegia from the baseline over a first 12-month period and a 12-month period of follow-up will be measured.

SECONDARY OUTCOMES:
Axial length change | Baseline, 1st year and 2nd year
  Axial length (mm) will be measured after cycloplegia using a non-contact optical biometer.
  Change in axial length from the baseline over a first 12-month period and a 12-month period of follow-up will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yan Yin Tse, PhD, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hon Y, Chun RKM, Leung TW, Qi H, Hasegawa K, Leung KY, To CH, Lam CSY, Tse DY. Myopia control efficacy of second-generation defocus incorporated multiple segments spectacle lenses on fast progressing myopes: Study protocol of a randomised controlled trial. PLoS One. 2025 Oct 31;20(10):e0335061. doi: 10.1371/journal.pone.0335061. eCollection 2025. PMID 41171741